CLINICAL TRIAL: NCT07206251
Title: The Effect of the Window Films on Cognition, Perception, and Health
Acronym: FOIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ERB2024BE34
Record Dates: First submitted 2025-03-20; First posted 2025-10-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Window Foil; Thermoregulation; Thermal Perception; Daylight; Saliva; Cognition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Windowed room (no foil added) (No Intervention): Regular Windowed room (no foil added)
- Foiled Windowed room (foil added) (Experimental): Foiled Windowed room (foil added)
  Interventions: Behavioral: Foiled Windowed room (foil added)

INTERVENTIONS:
Behavioral: Foiled Windowed room (foil added) — Foiled Windowed room (foil added)
  Arms: Foiled Windowed room (foil added)

SUMMARY:
To enable the Netherlands to reach the 2030 carbon emission goals, older homes need to be renovated to become more energy-efficient and comfortable. This project aims to provide shallow renovations of window films. These shallow renovations can be completed in 1-2 days and cost significantly less than a deep renovation. The study aims investigate how such window films can affect humans (low-e film and thermochromatic) if applicated in real life.

DETAILED DESCRIPTION:
This study consists of one screening session (1.5 hours) and two testing sessions (5.5 hours each)

Screening session:

In the screening session, a questionnaire about general information as well as a medical questionnaire that asks about, current health status, lifestyle, morningness-eveningness chronotype, use of contraceptives, and sleep quality are completed. This data is necessary to assess the eligibility and to analyse the collected data with consideration of possible effect of lifestyle.

Testing sessions:

Subjects will be exposed to 2 different conditions (window film vs. no window film) in two days (11:15- 16:45) to assess the window film(s) influence on visual and temperature comfort, sensation and perception. The exposure rooms are low-e film room (film 1) or a thermochromic film room (film 2), compared with no film room (control). These films will be applied to windows. 2 cognitive cognitive tests, 2 vision tasks and fill in questionanires at set times are performed. Also wearable sensors as mentiond in Part 3 section 2 to measure their physiological parametersm suchs as skin temperature, heart rate and physical activity. Lastly, every hour a saliva sample by spitting into a tube to measure the cortisol level in the saliva is provided. Saliva is collected to measure cortisol changes caused by the environment. The samples are then stored immediately in a -20 freezer, after it is transported to the storage lab they will be centrifuged for 2 mins at 1000g and then stored in a

-80 freezer for the duration of the study until analysis. The storage room is secured and only the research team can assess the samples. When the samples are to be analyzed for cortisol, the sample is defrosted and tested by a spectrophotometer to quantify the amount of cortisol. The sample is then discarded after this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Generally Healthy Adult
* Ages between 18-40 years old
* Normal or correct vision (with use of glasses or contact lenses)
* Full vision
* Both males or females

Exclusion Criteria:

* No Raynaud's syndrome
* No metabolic or cardiovascular diseases
* No ADHD or cognitive disorders
* No night shift work
* No colour blindness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Cognitive Performance Scores | 2 x in 5 hours test session both test days
  Participants completed 2 cognitive battery tests (Creyos) during each test day at 2 different timepoints; one early afternoon, the other late afternon.

SECONDARY OUTCOMES:
Skin Temperature | every 1 min it is collected automatically over 5 hours test day and 2 test days
  Temperature in celsius
Visual Scale | every 30mins to 1 hour over 5 hours test day and 2 sessions in total
  Visual perceptual likert scales

CONTACTS AND LOCATIONS:
Locations (1):
- Vertigo - TU/e, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No
Study is conducted by the researchers who will also process and analyse the data set anonymoously.